CLINICAL TRIAL: NCT05559957
Title: Isolated Oligohydramnios is Associated With Less Favorable Delivery and Composite Neonatal Outcomes
Brief Title: Isolated Oligohydramnios Less Favorable Delivery and Neonatal Outcomes
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hytham Atia, Associate professor, Zagazig University
Other Study IDs: AFHSRMREC/2020/OB/GYNAE/429
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Oligohydramnios, Delivered
MeSH Terms: conditions — Oligohydramnios

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Isolated oligohydramnios group: Cases with oligohydramnios (amniotic fluid index less than 5) without an overt underlying reason in the third trimester
  Interventions: Behavioral: observation of delivery and neonatal outcomes
- Normal amniotic fluid group: Normal pregnancy cases with normal amniotic fluid index
  Interventions: Behavioral: observation of delivery and neonatal outcomes

INTERVENTIONS:
Behavioral: observation of delivery and neonatal outcomes — MONITORING THE DELIVERY MODE EITHER CESAREAN OR VAGINAL, BESIDE THE NEONATAL OUTCOME AND MORBIDITIES IN BOTH GROUPS

SUMMARY:
Oligohydramnios happens in 1-5% of term pregnancies. The clinical significance of isolated oligohydramnios been a matter of debate. We aimed in this study to investigate the impact of isolated oligohydramnios on the mode of delivery and risk of adverse perinatal outcome.

DETAILED DESCRIPTION:
Retrospective study conducted in Armed Forces Hospitals of Southern Region, comparing cases with oligohydramnios (amniotic fluid level index <5) to normal amniotic fluid cases (amniotic fluid level index ≥ 8). Primary outcomes are the mode of delivery and adverse perinatal outcomes (including mortality, NICU admission, low Apgar score and sepsis)

ELIGIBILITY:
Inclusion Criteria:

1. Third trimester pregnancy
2. Isolated oligohydramnios

Exclusion Criteria:

1. Multiple pregnancy
2. less than 32 weeks
3. medical disorders like DM HPN
4. Fetal jeopardy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women between 32 and 41 weeks with otherwise normal pregnancy. Isolated oligohydramnios group are diagnosed with amniotic fluid index less than 5.
Sampling Method: Probability Sample
Enrollment: 636 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Delivery mode | through study completion, an average of 1 year
  Either vaginal delivery or cesarean section
Composite neonatal outcomes | through study completion, an average of 1 year
  Risk of low Apgar score, transient tachypnea of newborn, ICU admission, etc

SECONDARY OUTCOMES:
Induction of labor rate | through study completion, an average of 1 year
  Comparing incidence of labor induction between both groups and between gestational age groups

CONTACTS AND LOCATIONS:
Overall Officials: Hytham Atia Atia, M.D., Principal Investigator — Armed Forces Hospitals Southern Region KSA
Locations (1):
- Armed Forces Hospitals Southern Region, Khamis Mushait, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang J, Troendle J, Meikle S, Klebanoff MA, Rayburn WF. Isolated oligohydramnios is not associated with adverse perinatal outcomes. BJOG. 2004 Mar;111(3):220-5. doi: 10.1111/j.1471-0528.2004.00060.x. PMID 14961882